CLINICAL TRIAL: NCT01046721
Title: Investigation of the Cardiovascular Effects of Exenatide in Healthy Male Subjects
Brief Title: Study Looking at Cardiovascular Effects of Exenatide, Its Blood Pressure Lowering Effect and Its Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A/6/2009-exenatide-CVS
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
Keywords: blood pressure; superior mesenteric artery blood flow; cardiovascular effects; Exenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Active Comparator): subcutaneous administration of Exenatide (0.02ml)
  Interventions: Drug: Exenatide
- 0.9% Saline (Placebo Comparator): subcutaneous administration of 0.9% saline solution (0.02 ml)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Exenatide — single dose of 5 microg Exenatide. Subcutaneous administration
  Other Names: Byetta
  Arms: Exenatide
Drug: Saline — subcutaneous administration of 0.9% saline solution (0.02 ml)
  Other Names: 0.9% Saline solution
  Arms: 0.9% Saline

SUMMARY:
Exenatide is a new drug which lowers blood sugar (glucose) levels for people with type 2 diabetes. It has significant advantages over other treatments such as insulin as it causes weight loss in a group of people that is generally overweight. Data from studies involving exenatide have shown that it also has an effect on blood pressure. The mechanism for the blood pressure lowering effect is not known and has not been investigated previously. Exenatide may have an effect on blood vessels throughout the body and gut to reduce blood pressure. 12 healthy men (18-45yr) will be studied on 2 occasions. Limb blood flow, skin blood flow, gut blood flow, blood pressure, and heart rate will be measured half hourly for 4 hours. Blood samples (3ml) for insulin and glucose determination will be taken via a cannula and 3-way tap at the same time points. A dose of either 5μg exenatide or saline will be injected under the skin of the abdomen and a breakfast will be provided during the study. A urine collection will be made over the duration of the study.

DETAILED DESCRIPTION:
Background:

Glucagon-like peptide-1 (GLP-1) is an incretin hormone secreted from the L-cells of the gut following a meal (1). GLP-1 has multiple modes of action, including to augment the usual rise in insulin release and decrease in glucagon that follows carbohydrate ingestion (2). GLP-1 therefore plays a part in glucose homeostasis. GLP-1 secretion is reduced in patients with type 2 diabetes (T2DM) and extended-action GLP-1 agonists or mimetics are currently being introduced for use as glucose lowering medications. The peptide exendin-4 has considerable homology with GLP-1 but is resistant to degradation by the enzyme Dipeptidyl peptidase-4 (DPP-IV) and so has a much longer duration of action. The synthetic exendin, 'Exenatide', is a novel GLP-1 mimetic which has recently been licensed for the treatment for T2DM and has shown to be an effective glucoregulatory agent when administered as a twice- daily subcutaneous injection (11).

GLP-1 agonists give a low risk of significant hypoglycaemia as effects on insulin and glucagon are largely glucose-dependent. In addition, considerable weight loss is often observed with GLP-1 agonists in clinical practice, and these drugs are currently being considered in treating obesity, even outside the context of diabetes.

A moderate blood-pressure (BP) lowering effect of GLP-1 agonists has also been noted as a secondary outcome measure in large clinical trials in patients with T2DM. In one such study, Exenatide was associated with a reduction in systolic/diastolic BP of 5/2 mmHg The mechanism for this apparent hypotensive effect is not known. An infusion of GLP-1 agonists induces a natriuresis, which may contribute to a reduction in BP.

Aims:

The aim of this study is to assess the cardiovascular effects of Exenatide in young, healthy, non-obese male subjects. We propose to compare the effect of Exenatide vs. placebo and study the cardiovascular effects by a number of non invasive techniques.

Experimental protocol and methods:

12 healthy male subjects aged 18-45 years with BMI 20-27 kg/m2 will be recruited. Subjects will attend for an initial screening visit and initial assessments. This will enable familiarization with the room and equipment to be used. On arrival at the laboratory, subjects will be asked to void their bladder and a urine collection will be commenced. Subjects will be asked to wear shorts during the study and rest semi-supine on a hospital bed. They will place their hand in a heated hand warming unit and an intravenous cannula will be inserted, for arterialized venous blood sampling,. Subjects will rest for 1hour before receiving either Exenatide or placebo injection. Measurements of Limb blood flow (by venous occlusion plethysmography); skin blood flow (by laser Doppler); blood pressure, heart rate (HR) and cardiac output (by Finometry™);and regional blood flow (by ultrasound imaging and flow velocity measurement of the superior mesenteric arteries (SMA) will take place every 30minutes. Blood sampling for insulin and glucose will be carried out every 15minutes throughout the study. Subjects will rest for 120 minutes after injection with measurements every 30 minutes as before with blood sampling every 15 minutes until 120 minutes post injection. Subjects will receive a high carbohydrate breakfast 60 minutes post injection. Urine will be collected during the study to assess urinary sodium excretion.

Measurable end points/statistical power of the study:

Our primary end point will be to measure meal induced changes in superior mesenteric (SMA) blood flow in the 2 groups (Exenatide vs. placebo.)Secondary endpoints will be measures including: BP, HR, Limb Blood Flow, Skin Blood Flow, and peripheral resistance responses when fasted and after eating- (both Exenatide and placebo groups).

From previous studies we calculated that SMA blood flow at rest = 346 (27) ml/min and peak SMA blood flow after high carbohydrate meal = 611(80) ml/min. With 12 subjects, a reduction in blood flow of 71ml/min, following Exenatide injection, would be required if powered at 80%.

ELIGIBILITY:
Inclusion Criteria:

* male,
* non-obese (BMI 20-27: those with a BMI > 25 will be excluded if they have a waist circumference > 90cm),
* aged 18-45yrs,
* non-smoker.

Exclusion Criteria:

* any metabolic or endocrine abnormalities,
* clinically significant abnormalities on screening,
* taking regular medication.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
superior mesenteric (SMA) blood flow | 0, 30, 60, 90, 120, 150, & 180 min after meal
  Meal induced changes in superior mesenteric (SMA) blood flow - exenatide versus placebo.

SECONDARY OUTCOMES:
Blood Pressure (BP) | 0, 30, 60, 90, 120, 150, & 180 min after meal
  BP responses when fasted and after eating- Exenatide vs. placebo.
Heart Rate (HR) | 0, 30, 60, 90, 120, 150, & 180 min after meal
  HR responses when fasted and after eating- Exenatide vs. placebo.
Limb Blood Flow (LBF) | 0, 30, 60, 90, 120, 150, & 180 min after meal
  Limb Blood Flow responses when fasted and after eating- Exenatide vs. placebo.
Skin Blood Flow | 0, 30, 60, 90, 120, 150, & 180 min after meal
  Skin Blood Flow responses when fasted and after eating- Exenatide vs. placebo.
Peripheral resistance | 0, 30, 60, 90, 120, 150, & 180 min after meal
  peripheral resistance responses when fasted and after eating- Exenatide vs. placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Peter I Mansell, FRCP, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Laboratories, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendis B, Simpson E, MacDonald I, Mansell P. Investigation of the haemodynamic effects of exenatide in healthy male subjects. Br J Clin Pharmacol. 2012 Sep;74(3):437-44. doi: 10.1111/j.1365-2125.2012.04214.x. PMID 22320349